CLINICAL TRIAL: NCT00825721
Title: A Randomized, Placebo-Controlled, Single-Masked, Dose-Ranging Study of C-KAD Ophthalmic Solution in Patients With Loss of Visual Function Due to Age-Related Nuclear Cataracts
Brief Title: Dose-Ranging Study of an Ophthalamic Solution in Patients With Loss of Visual Function Due to Age-Related Nuclear Cataract
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chakshu Research, Inc. (Industry)
Responsible Party: Watiri Kamau-Kelley /Manager, Clinical & Regulatory Affairs, Chakshu Reserach, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CK-0105
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Nuclear Cataract
Keywords: Cataract Study; Ophthalmic Study; Agerelated cataract; Nuclear Cataract; Low grade nuclear cataracts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.3% (low dose) (Active Comparator)
  Interventions: Drug: C-KAD Ophthalmic Solution
- 2% (medium dose) (Active Comparator)
  Interventions: Drug: C-KAD Ophthalmic Solution
- 2.6% (high dose) (Active Comparator)
  Interventions: Drug: C-KAD Ophthalmic Solution
- Placebo (Placebo Comparator)
  Interventions: Drug: LiquiTears

INTERVENTIONS:
Drug: LiquiTears — 4 drops applied daily for 360 days
  Arms: Placebo
Drug: C-KAD Ophthalmic Solution — 4 drops applied daily for 360 days
  Arms: 1.3% (low dose)
Drug: C-KAD Ophthalmic Solution — 4 drops applied daily for 360 days
  Arms: 2% (medium dose)
Drug: C-KAD Ophthalmic Solution — 4 drops applied daily for 360 days
  Arms: 2.6% (high dose)

SUMMARY:
This study will evaluate the safety and efficacy of three doses of C-KAD Ophthalmic Solution in patients with loss of visual function due to age-related nuclear cataract

ELIGIBILITY:
Inclusion Criteria:

* Presence of nuclear sclerosis cataract
* BCDVA within the range of 20/40 and 20/80

Exclusion Criteria:

* Any other clinical condition in the eye that may compromise vision
* Presence or history of glaucoma
* Presence or history of diabetes
* Use of eyedrops
* Use of steroids

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-11; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity by ETDRS | 360 days

CONTACTS AND LOCATIONS:
Overall Officials: Sanduk Ruit, MD, Principal Investigator — Tilganga Eye Center; Reeta Gurung, MD, Principal Investigator — Tilganga Eye Center
Locations (1):
- Tilganga Eye Center, Kathmandu, Kathmandu, Nepal